CLINICAL TRIAL: NCT04179695
Title: Optimizing PD Patient's Health Pathways: Favoring Global, Patient Centered Care by a New Communication Aid Tool PARKINSUN
Brief Title: Evaluation of a New Communication Aid Tool to Favor Global Patient Centered Care
Acronym: PARKINSUN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Expert center of Parkinson's Disease (CHU Lille) (Unknown); College of teaching general practitioners (CEMG Lille) (Unknown); Regional Health Agency (ARS) (Unknown); UCB Pharma (Industry); Orkyn' (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018_74; 2019-A01008-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease
Keywords: Health pathway; patient centered care; communication aid- tool; primary care; secondary care
MeSH Terms: conditions — Parkinson Disease | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- consultation with Parkinsun (Experimental)
  Interventions: Other: Consulting with PARKINSUN as communication aid-tool
- consultation as usual without Parkinsun (Active Comparator)
  Interventions: Other: Consulting without PARKINSUN as communication aid-tool

INTERVENTIONS:
Other: Consulting with PARKINSUN as communication aid-tool — Participating patients visit their general practitioner or neurologist with PARKINSUN at 1 months, 4 months, 7 months
  Arms: consultation with Parkinsun
Other: Consulting without PARKINSUN as communication aid-tool — Participating patients visit their general practitioner or neurologist without PARKINSUN at 1 months, 4 months, 7 months
  Arms: consultation as usual without Parkinsun

SUMMARY:
PARKINSUN is a new communication aid tool, expected to favor global patient centered care for PD patients during consultation with GPs and neurologists. Two groups of patients will be randomized to use or not PARKINSUN when they consult their physicians every 3 months during 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women with all stages of PD
* Without severe chronic neurological or mental or psychiatric pathology
* Absence of cognitive impairment affecting autonomy (MDS criteria of dementia and MOCA > 22)
* able to come (alone or accompanied) to consultation
* Affiliate or beneficiary of a social security scheme
* Subject having signed informed consent
* Patient willing to comply with all procedures of the study and its duration

Exclusion Criteria:

* Administrative reasons: impossibility of receiving informed information, inability to participate in the whole study, absence of coverage by the social security system, refusal to sign consent.
* Subject under tutelage or curtailer.
* Subject not fluent in the French language to understand the instructions necessary to carry out the cognitive tests.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
variation of the delta of G-MISS Questionnaire | at 7 months

SECONDARY OUTCOMES:
G-MISS-Questionnaire at the end of each consultation (1 month, 4 months and 7 months) | at the end of each consultation (1 month and 7 months)
  Patient's satisfaction will be assessed by the G-MISS-Questionnaire. The G-MISS questionnaire is a standardized and validated tool in French. This questionnaire is taken from the American MISS-21 questionnaire, already used in neurologists to measure the satisfaction of patients with PD, after consultation It is easy to use with an average filling time of 6 minutes.
Global score of PARKINSUN | at the end of each consultation ((1 month and 7 months)
Individuals scores of PARKINSUN | at the end of each consultation ((1 month and 7 months)
MDS-UPDRS scores | at the end of each consultation ((1 month and 7 months)
PDQ-39 scores 6. Interpersonal Reactivity Index (IRI) | at the end of each consultation ((1 month and 7 months)
Likert Scale | at the end of each consultation (1 month and 7 months)
Interpersonal Reactivity Index (IRI) | at the end of each consultation (1 month and 7 months)

CONTACTS AND LOCATIONS:
Overall Officials: David Devos, Principal Investigator — University Hospital, Lille
Locations (1):
- Hopital Roger Salengro, CHU Lille, Lille, France